CLINICAL TRIAL: NCT04796545
Title: A Prospective, Multicenter Post-marketing Clinical Investigation of the SING IMT(TM) System, Model NG SI IMT 3X in Patients With Central Vision Impairment Associated With End-stage Age-related Macular Degeneration
Brief Title: Post-market Clinical Investigation of the SING IMT System, Model NG SI IMT 3X in Patients With End-stage Age-related Macular Degeneration
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: VisionCare, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: SING IMT PMCF
Record Dates: First submitted 2021-03-03; First posted 2021-03-15 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2025-11

CONDITIONS: AMD; Age-Related Macular Degeneration
Keywords: Age Related Macular Degeneration; Dry AMD; End-stage age-related macular degeneration; Central vision impairment; Geographic atrophy
MeSH Terms: conditions — Macular Degeneration; Geographic Atrophy | interventions — Drug Delivery Systems

STUDY DESIGN:
Intervention Model Description: SING IMT(TM) System, model NG SI IMT 3X
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- SING IMT System model NG SI IMT 3X (Experimental): All participants will be implanted with the SING IMT System model NG SI IMT 3X.
  Interventions: Device: SING IMT(TM) System, model NG SI IMT 3X

INTERVENTIONS:
Device: SING IMT(TM) System, model NG SI IMT 3X — The SING IMT 3X implant is a visual prosthetic implantable device, which, when combined with the optics of the cornea, constitutes a telephoto system for improvement of visual acuity in patients with bilateral, end-stage age-related macular degeneration.

SUMMARY:
The objective of this study is to demonstrate the safety and effectiveness of the SING IMT (Smaller Incision New Generation Implantable Miniature Telescope) 3X implant in improving vision in patients with central vision impairment associated with end-stage Age-related Macular Degeneration (AMD).

Eligible patients will be implanted with the SING IMT device and will be followed-up for a period of 12-months with post-operative ophthalmic exams and low-vision rehabilitation sessions.

DETAILED DESCRIPTION:
This is an interventional, prospective, multicenter, open label, single group assignment Post-Market Clinical Follow-up (PMCF) study in men and women >=55 years with central vision impairment associated with end-stage AMD.

Following completion of informed consent, patients will be evaluated for eligibility to enroll into the study. Baseline visual acuity of the study subjects will be assessed with a 2.8X external telescope simulator (ETS) using Early Treatment Diabetic Retinopathy Study (ETDRS) charts to determine if they are likely to benefit from receiving the IMT. To be included in the study and to proceed with the surgery, subjects must achieve, using the ETS, at least a one line (5 or more letters) improvement in distance on the ETDRS chart in the eye scheduled for surgery. Subjects not meeting these criteria will be excluded from the study.

If eligible, they will be scheduled for out-patient surgery to implant the IMT during routine cataract surgery.

Postoperatively, the surgeon will complete a usability and satisfaction questionnaire after each implantation procedure.

The patients will undergo ophthalmic evaluations in both eyes at regular intervals for up to 12 months. The subjects will also be required to undergo 6 to 10 additional visits for vision training with a low vision specialist.

Surgical complications, as well as all Adverse Event (AEs) and use of medications will be monitored from baseline to the end of the study.

ELIGIBILITY:
Inclusion Criteria:

1. Be 55 years of age or older.
2. Have retinal findings of geographic atrophy or disciform scar with foveal involvement as determined by fluorescein angiography or OCT.
3. Have evidence of cataract.
4. Have best-corrected distance visual acuity (BCDVA) no better than 20/80 (0.6 LogMAR) and no worse than 20/800 (1.6 LogMAR) in both eyes.
5. Have adequate peripheral vision in the eye not scheduled for surgery, assessed by observation of ambulation.
6. Achieve at least a five-letter improvement on the ETDRS chart in the eye scheduled for surgery when using Samsara's 2.8X external telescope simulator (ETS, supplied separately).
7. Have an ACD of at least 2.5 mm in the eye scheduled for surgery.
8. Be willing to participate in a post-operative training program for the use of the NG SI IMT 3X implant.
9. Review and sign the Independent Ethics Committee (IEC)-approved Informed Consent Form (ICF) prior to any study-related procedures being performed.
10. Have adequate understanding of the local language to understand verbal and written subject information and be willing to comply with the study requirements.

Exclusion Criteria:

1. Evidence of active choroidal neovascularization (CNV) on fluorescein angiography or OCT or were treated for CNV within the past six months.
2. Any ophthalmic pathology that compromises the patient's peripheral vision in the fellow eye.
3. A history of steroid-responsive rise in IOP, uncontrolled glaucoma, or preoperative IOP>22 mm Hg.
4. Corneal guttata.
5. Known sensitivity to post-operative medications.
6. Significant communication impairment or severe neurological disorders.
7. Have undergone previous intraocular or corneal surgery of any kind in the operative eye, including any type of surgery for either refractive or therapeutic purposes.
8. An ocular condition that predisposes the patient to eye rubbing.
9. Prior or expected ophthalmic-related surgery within 30 days preceding the NG SI IMT 3X implant surgery.
10. Patients for whom the planned operative eye has:

    * Myopia > 6.0 D
    * Hyperopia > 4.0 D
    * Axial length < 21 mm
    * Endothelial cell density < 1600 cells per square mm
    * Narrow angle, i.e., < Schaffer grade 2.
11. Inflammatory ocular disease.
12. Cornea stromal or endothelial dystrophies, including guttata.
13. Zonular weakness/instability of crystalline lens, or pseudoexfoliation.
14. Diabetic retinopathy.
15. Untreated retinal tears.
16. Retinal vascular disease.
17. Optic nerve disease.
18. A history of retinal detachment.
19. Retinitis pigmentosa.
20. Intraocular tumor.
21. Have received any investigational product within 30 days prior to study enrollment or be planning to participate in another investigation during the course of this study.
22. Be an employee (or a relative of an employee) of the contract research organization (CRO) responsible for conducting the study, Sponsor, or Sponsor representative.
23. Have a condition or be in a situation that, in the Investigator's opinion, may put the Subject at significant risk, may confound the study results, or may interfere significantly with the Subject's participation in the study.

Min Age: 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 76 (Estimated)
Dates: Start 2022-09-13 (Actual); Primary Completion 2027-02 (Estimated); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
Safety of the SING IMT System, model NG SI IMT 3X, including its delivery system | 12 months
  The percent decrease in endothelial cell density (ECD).

SECONDARY OUTCOMES:
Incision size needed for device implantation | 12 moths
  Incision size will not exceed 8.0 mm (non-inferiority assumption) in 75% of surgeries
Surgical complications | 12 moths
  AEs and serious adverse events
Improvement in near and distance best corrected visual acuity (BCVA) in implanted eyes. | 12 months
  Near and distance BCVA will show an improvement of ≥2 lines in the ETDRS chart in at least 50% (non-inferior to 50%) of the implanted eyes at 12 months post implantation.
Usability of SING IMT System, including delivery system | 12 months
  Surgeon will complete a usability and satisfaction questionnaire

OTHER OUTCOMES:
Device stability and fixation | 12 months
  Assessed by slit lamp biomicroscopy examination: device tilt and device decentration
Post-operative anterior chamber depth (ACD) | 12 months
  Anterior Chamber Depth (ACD) evaluated by ultrasound biomicroscopy (UBM), ocular coherence tomography (OCT) or another applicable test method

CONTACTS AND LOCATIONS:
Locations (13):
- UZ Brussel, Brussels, Belgium
- France (3):
  - Centre d'Ophtalmologie Paradis-Monticelli, Marseille
  - Hélios Ophtalmologie, Saint-Jean-de-Luz, Saint-Jean-de-Luz
  - CHRU de Strasbourg, Strasbourg
- Germany (2):
  - Augenklinik Städtisches Klinikum Karlsruhe, Karlsruhe
  - Universitätsklinikum Münster Klinik für Augenheilkunde, Münster
- Mater Misericordiae University Hospital, Dublin, Ireland
- Italy (2):
  - Università degli Studi di Napoli Federico II, Napoli
  - Fondazione Policlinico Universitario Agostino Gemelli, Roma
- Spain (3):
  - VISSUM, Alicante
  - Institut OMIQ, Barcelona
  - Hospital Universitario La Luz - Quirónsalud, Madrid
- Royal Victoria Hospital Belfast Health & Social Care Trust, Belfast, United Kingdom

IPD SHARING:
Plan to Share IPD: No